CLINICAL TRIAL: NCT06635122
Title: Case-Control Study of Transjugular Intrahepatic Portosystemic Shunt in Treating Platinum-Related Porto-Sinusoidal Vascular Disease With Esophagogastric Variceal Bleeding
Brief Title: TIPS for Platinum-Related Porto-Sinusoidal Vascular Disease With Variceal Bleeding
Status: Active, not recruiting | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tie Jun, Director of clinical research, Air Force Military Medical University, China
Other Study IDs: KY20242274-C-1
Record Dates: First submitted 2024-10-05; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Porto-Sinusoidal Vascular Disease; Cirrhosis Due to Hepatitis B; Esophageal Variceal Rebleeding; Gastric Variceal Bleeding
MeSH Terms: conditions — Idiopathic Noncirrhotic Portal Hypertension | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental group: TIPS for PSVD: This group of PSVD patients received TIPS treatment.TIPS is an artificial channel within the liver that establishes communication between the inflow portal vein and the outflow hepatic vein.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt
- Control group: Endoscopic therapy for PSVD: This group of PSVD patients received endoscopic treatment.Endoscopic treatment includes endoscopic variceal ligation, endoscopic injection sclerotherapy and endoscopic variceal histoacryl injection therapy
  Interventions: Procedure: Endoscopic treatment
- Control Group: TIPS for Cirrhosis Due to Hepatitis B: This group of Cirrhosis Due to Hepatitis B patients received TIPS treatment.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt — Transjugular intrahepatic portosystemic shunt (TIPS) is a procedure that uses imaging guidance to connect the portal vein to the hepatic vein in the liver. The TIPS-dedicated stent (Gore, Arizona, USA)was emplaced within the liver and gradually expanded utilizing a balloon with a diameter ranging from 6 to 10 millimeters, aiming for a decrease in portal-venous pressure gradient to less than 12 mmHg or achieve a reduction of 25 to 50% relative to the baseline pressure.
  Groups: Control Group: TIPS for Cirrhosis Due to Hepatitis B; Experimental group: TIPS for PSVD
Procedure: Endoscopic treatment — Endoscopic variceal ligation, endoscopic injection sclerotherapy, endoscopic variceal histoacryl injection therapy , or a combination of several methods were selected according to the location, size, and shape of the patient's varicose veins.Treatment failure can be transferred to TIPS therapy.
  Groups: Control group: Endoscopic therapy for PSVD

SUMMARY:
Platinum-based compounds are associated with several adverse effects, including Porto-Sinusoidal Vascular Disease (PSVD). Therapeutic strategies for platinum-related PSVD are based on the management of complications seen in cirrhotic portal hypertension. Currently, a combination of non-selective beta-blockers (NSBB) and endoscopic therapies, such as endoscopic band ligation and endoscopic cyanoacrylate injection, is recommended as the primary approach for the secondary prevention of variceal rebleeding, with Transjugular Intrahepatic Portosystemic Shunt (TIPS) reserved for cases in which first-line treatments fail.

However, previous research indicates that endoscopic treatments for the secondary prevention of esophagogastric variceal bleeding show suboptimal efficacy in PSVD patients. In contrast, TIPS has demonstrated comparable rebleeding control but with a lower incidence of liver-related complications and reduced mortality in PSVD patients compared to cirrhotic patients with similar liver function. Based on these findings, the investigators hypothesize that TIPS may be a safer option for this cohort, offering lower rebleeding rates than endoscopic therapy, reduced incidences of hepatic encephalopathy and liver insufficiency, and improved survival rates compared to patients with cirrhosis.

DETAILED DESCRIPTION:
Platinum-based compounds are widely employed in chemotherapy regimens, yet they are associated with a range of adverse effects, most notably Porto-Sinusoidal Vascular Disease (PSVD). PSVD can trigger portal hypertensive complications, including esophagogastric varices and ascites.

Platinum-related PSVD constitutes a variant of intrahepatic presinusoidal portal hypertension, manifesting clinical symptoms analogous to those of liver cirrhosis. There is a scarcity of clinical data pertaining to these patients, and therapeutic strategies should be extrapolated from the management of complications associated with cirrhotic portal hypertension. Presently, the combination of non-selective beta-blockers (NSBB) with endoscopic therapies is advocated as the primary therapeutic modality for the secondary prevention of variceal bleeding, with transjugular intrahepatic portosystemic shunt (TIPS) being employed subsequent to the failure of firstline treatments.

A study by Shanghai Zhongshan Hospital revealed that patients with gastroesophageal variceal bleeding following oxaliplatin-based chemotherapy required more frequent endoscopic treatments to prevent rebleeding compared to those with cirrhosis, and exhibited higher rates of rebleeding and mortality. This suggests the suboptimal efficacy of endoscopic treatments for secondary prevention in this patient population. Additionally, findings from a retrospective study conducted by our institution demonstrated that PSVD patients treated with TIPS for variceal bleeding achieved rebleeding control comparable to cirrhotic patients with similar liver function. However, PSVD patients experienced a lower incidence of liver-related complications, such as overt hepatic encephalopathy and hepatic insufficiency, along with a reduced mortality rate.

Therefore, it is postulated that patients with platinum-related PSVD and esophagogastric varices may experience a lower rebleeding rate following TIPS intervention compared to those receiving endoscopic treatment, without an increased risk of hepatic encephalopathy. TIPS may present a safer treatment option for this cohort, with a reduced incidence of hepatic encephalopathy and liver insufficiency, and improved survival rates compared to patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years and confirmed diagnosis of Platinum-Related Porto-Sinusoidal Vascular Disease or Cirrhosis Due to Hepatitis B
* Acute esophagogastric variceal bleeding or history of gastroesophageal variceal bleeding episodes
* The patients was received endoscopic variceal ligation/histoacryl injection therapy or TIPS treatment
* At least one postoperative follow-up data

Exclusion Criteria:

* Primary tumor recurrence and metastasis
* Hepatocellular carcinoma or other malignant tumors
* Common contraindications of TIPS
* HIV, AIDS, Serious acute and chronic disease
* Pregnant or breast-feeding woman
* Without postoperative follow-up data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients confirmed diagnosis of Platinum-Related Porto-Sinusoidal Vascular Disease or Cirrhosis Due to Hepatitis B in Xijing Hospital and Shanghai Zhongshan Hospital during Jan 2010 to Jun 2024
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of clinically significant variceal rebleeding | 12 months
  Recurrent melena or hematemesis resulting in either hospital admission, blood transfusion, drop in hemoglobin of at least 3 g/L, or death within 6 weeks after rebleeding.

SECONDARY OUTCOMES:
Cumulative incidence of death | 12 months
  all cause mortality
Cumulative incidence of hepatic encephalopathy (HE) | 12 months
  HE is classified as covert HE and overt HE
Cumulative incidence of patients with other decompensation events | 12 months
  Decompensation was defined as hepatic ascites, abdominal ascites jaundice and infection
Cumulative incidence of liver function damage | 12 months
Cumulative incidence of treatment related complications | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tie, M.D.,Ph.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided